PATIENT INFORMATION SHEET / POSSIBLE PARTICIPANT

TITLE OF THE STUDY: BARIATRIC SURGERY IN PATIENTS WITH

SCHIZOPHRENIA

STUDY CODE: IIBSP-BAR-2022-30

**PROMOTER:** Sant Pau Hospital Research Institute la Santa Creu– IIB Sant Pau

PRINCIPAL INVESTIGATOR: Inka Miñambres, Endocrinology and Nutrition

Service. Phone 935565661

CENTRE: Hospital de la Santa Creu i Sant Pau.

INTRODUCTION

We are writing to inform you about a research study in which you are invited to participate.

The study has been approved by the corresponding Clinical Research Ethics Committee.

Our intention is only that you receive the correct and sufficient information so that you can

evaluate and judge whether or not you want to participate in this study. To do this, read this

information sheet carefully and we will clarify any doubts that may arise after the explanation.

In addition, you can consult with the people you consider appropriate.

VOLUNTARY PARTICIPATION

You should know that your participation in this study is voluntary and that you can decide

not to participate or change your decision and withdraw your consent at any time, without

altering your relationship with your doctor or affecting your treatment.

GENERAL DESCRIPTION OF THE STUDY

It is known that schizophrenia is associated with obesity in a significant number of

patients and it implies a poor prognostic factor, with weight loss being important in this

population. However, data about the prognosis of weight loss surgery in subjects with

schizophrenia is scant. The objective of this study is to retrospectively analyze the cases of

patients with schizophrenia (study group) who have undergone weight loss surgery with the

Study code:

Version: 2. Date: 06/02/2022

1

intention of analyzing the beneficial effects of the surgery, as well as the complications. in

this group of patients. In parallel, the data of patients who do not suffer from any psychiatric

illness (control group) will be collected. You will be invited to participate as a study group

or as a control group depending on your characteristics.

As it is a retrospective data collection, the study does not require additional visits or tests to

the usual ones and does not entail any additional risk for the patient. No adverse effects are

anticipated as no procedure will be performed.

The total number of patients expected to be included in the study will be 20 patients and 80

controls aproximately

BENEFITS AND RISKS DERIVED FROM YOUR PARTICIPATION IN THE

**STUDY** 

It is likely that the present study does not result in a direct benefit on the health of the subjects

participating in the study. However, it is intended to expand knowledge about the prognosis

of weight reduction surgery in subjects with schizophrenia and this knowledge may in the

future improve the selection of which cases should undergo bariatric surgery and which cases

the risks of surgery would outweigh the benefits. .

CONFIDENTIALITY

The treatment, communication and transfer of personal data of all participating subjects will

comply with the provisions of Regulation (EU) No. 2016/679 and Organic Law 3/2018, of

December 5, Protection of Personal Data and Guarantee of Digital Rights.

Both the Center and the Promoter are respectively responsible for the processing of your data

and undertake to comply with the data protection regulations in force. The data collected for

the study will be identified by a code and only your study doctor/collaborators will be able to

associate said data with you and your medical history. Therefore, your identity will not be

disclosed to any person, except for exceptions, in case of medical emergency or legal

requirement.

Access to your personal information will be restricted to the study doctor/collaborators, health

authorities, the Research Ethics Committee and personnel authorized by the sponsor (study

Study code:

Version: 2. Date: 06/02/2022

2

monitors, auditors), when needed to verify the study data and procedures, but always

maintaining their confidentiality in accordance with current legislation.

In accordance with the provisions of the data protection legislation, you can exercise the rights

of access, modification, opposition and cancellation of data. You can also limit the processing

of data that is incorrect, request a copy or transfer to a third party (portability) the data that

you have provided for the study. To exercise your rights, you can contact the main researcher

of the study. You can also exercise your rights by sending a written communication to the

following address: c/Sant Quintí 77-79 08041 Barcelona. Likewise, you have the right to

contact the Data Protection Agency if you are not satisfied.

If you decide to withdraw consent to participate in this study, no new data will be added to

the database. However, you should note that the data cannot be deleted even if you stop

participating in the study, to ensure the validity of the research and to comply with legal

duties.

The investigator and the sponsor are obliged to keep the data collected for the study for at

least 5 years after its completion. Subsequently, your personal information will only be kept

by the health care center and by the sponsor for other scientific research purposes if you have

given your consent to do so, or if permitted by law and applicable ethical requirements.

If we transfer your encrypted data outside the EU to our group entities, service providers

or scientific researchers who collaborate with us, the participant's data will be protected

with safeguards such as contracts or other mechanisms by data protection authorities.

data. If the participant wants to know more about it, they can contact the Principal

Investigator of the study or the Promoter's Data Protection Officer by email at

dpo ir@santpau.cat.

**ECONOMIC COMPENSATION** 

Your participation in the study will not entail any expense or financial compensation. You

will not have to pay for the study procedures.

OTHER RELEVANT INFORMATION

Study code:

Version: 2. Date: 06/02/2022

3

If you choose to withdraw consent to participate in this study, no new data will be added to the database and you may require the destruction of all identifiable samples previously withheld to prevent further testing.

By signing the attached consent form, you agree to abide by the study procedures that have been disclosed to you.

If you have any questions or want more information, you can contact the principal investigator of the study.

Thank you very much for your help.

## **INFORMED CONSENT**

Study title: BARIATRIC SURGERY IN PATIENTS WITH SCHIZOPHRENIA

| I (first and last name) |
|--------------------------------------------------------------|
| I have read the information sheet that has been given to me. |
| I have been able to ask questions about the study. |
| I have received enough information about the study. |
| I have spoken with: |
| (first and last name of the researcher) |
| I understand that my participation is voluntary. |
| I understand that I can withdraw from the study: |

1° Whenever I want

2° Without having to give explanations.

3° Without this affecting my medical care.

Study code: 4

Version: 2. Date: 06/02/2022

Patient's signature **Investigator Signature** Date: Date: This document will be signed in duplicate, keeping one copy for the researcher and another for the patient. INFORMED CONSENT Study title: BARIATRIC SURGERY IN PATIENTS WITH **SCHIZOPHRENIA** I (name and surname) ......in the capacity of.....(relationship with the participant) of..... .....(name and surname of the participant) I have read the information sheet that has been given to me. I have been able to ask questions about the study. I have received enough information about the study. I have spoken with: (first and last name of the researcher) I understand that patient participation is voluntary. I understand that I can withdraw from the study: 1° Whenever I want 2° Without having to give explanations.

- I freely give my consent to participate in the study and give my consent for the access

and use of my data under the conditions detailed in the information sheet.

Study code: 5

Version: 2. Date: 06/02/2022

| 3° Without this affecting your me | edical care. |
|---|---|
| - In my presence, | (name of participant) has been |
| given all relevant information ad | apted to their level of understanding and they agree to |
| participate. I give my consent for | (name of participant) to |
| participate in this study and I giv | ve my consent for the access and use of the data under |
| the conditions detailed in the info | ormation sheet. |
| Signature of representative | Signature of investigator |
| Date : | Date : |
| N. C. O. | MED CONCENT |
| INFOR | MED CONSENT |
| Study title: BARIATRIC SURGER | Y IN PATIENTS WITH |
| SCHIZOPHRENIA | |
| [( | name and surname of the witness) declare under my |
| own responsibility that | (name and surname of the |
| participant) | |
| You have read (or it has been read to yo | ou, in the case in which the patient cannot read), the |
| nformation sheet that has been given to yo | ou. |
| You have been able to ask questi | ons about the study. |
| You have received enough inform | nation about the study. |
| Has spoken with: | |
| (first and last name of the research | shor) |
| thist and last name of the researc | |

Study code: 6

Study code: Version: 2. Date: 06/02/2022 You understand that your participation is voluntary.

You understand that you can withdraw from the study:

- 1° Whenever I want
- 2° Without having to give explanations.
- 3° Without this affecting your medical care.
- You have freely expressed your agreement to participate in this study and give your consent for the access and use of the data under the conditions detailed in the information sheet.

| Witness signature | Investigator Signature |
|-------------------|------------------------|
| Date : | Date : |

This document will be signed in duplicate, keeping one copy for the researcher and another for the patient.

Study code: 7

Version: 2. Date: 06/02/2022